CLINICAL TRIAL: NCT07242729
Title: Bone Marrow Aspirate Versus Platelet-Rich Fibrin for the Treatment of Plantar Fasciitis - A Double-Blind Randomized Clinical Trial
Brief Title: Bone Marrow Aspirate Versus Platelet-Rich Fibrin for the Treatment of Chronic Plantar Fasciitis
Acronym: fasciitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rodrigo de Almeida Mastrorosa, Principal Investigator / PhD Candidate, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 90411925.0.0000.5505
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Plantar Fasciitis
Keywords: Plantar Fasciitis; Bone Marrow Aspirate; Platelet-Rich Fibrin; Ultrasound-Guided Injection; Regenerative Medicine
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel, randomized, controlled clinical trial comparing the effects of ultrasound-guided injection of Bone Marrow Aspirate versus Platelet-Rich Fibrin in patients with chronic plantar fasciitis.
Who Masked: Participant, Investigator
Masking Description: Double-blind design: both participants and investigators performing follow-up assessments are blinded to group allocation. The injectate is prepared in a separate room by a technician not involved in patient assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone Marrow Aspirate (BMA) Group (Experimental): Participants receive a single ultrasound-guided injection of autologous bone marrow aspirate (approximately 8 mL) into/around the plantar fascia on one side, according to randomization.
  Bone marrow aspirate is obtained from the posterosuperior iliac crest under local anesthesia and prepared under sterile conditions. The injection is performed after regional anesthesia of the tibial nerve using ultrasound guidance.
  Interventions: Biological: Bone Marrow Aspirate Injection
- Platelet-Rich Fibrin (PRF) Group (Experimental): Participants receive a single ultrasound-guided injection of autologous platelet-rich fibrin (PRF, approximately 8 mL) into/around the plantar fascia on the contralateral side, according to randomization.
  PRF is prepared from 60 mL of venous blood centrifuged without anticoagulant to form a fibrin clot, which is injected into the painful area of the fascia after regional anesthesia of the tibial nerve under ultrasound guidance.
  Interventions: Biological: Platelet-Rich Fibrin Injection

INTERVENTIONS:
Biological: Bone Marrow Aspirate Injection — Ultrasound-guided injection of autologous bone marrow aspirate obtained from the posterosuperior iliac crest under local anesthesia. Approximately 8mL of aspirate is injected into/around the plantar fascia.
  Other Names: BMA
  Arms: Bone Marrow Aspirate (BMA) Group
Biological: Platelet-Rich Fibrin Injection — Ultrasound-guided injection of autologous platelet-rich fibrin (PRF) prepared from 60 mL of venous blood centrifuged to form a fibrin clot. Approximately 8mL of PRF is injected into/around the plantar fascia.
  Other Names: PRF
  Arms: Platelet-Rich Fibrin (PRF) Group

SUMMARY:
This randomized, double-blind clinical trial aims to compare the clinical and imaging effects of autologous bone marrow aspirate versus platelet-rich fibrin injections in patients with chronic plantar fasciitis. The procedures are performed under ultrasound guidance to ensure precision and safety. The study evaluates pain reduction, foot function, and ultrasonographic changes in the plantar fascia at follow-up intervals.

DETAILED DESCRIPTION:
Chronic plantar fasciitis is a common cause of heel pain that may persist despite standard conservative measures such as physical therapy, stretching, orthoses, and corticosteroid injections. Regenerative medicine techniques, including autologous platelet concentrates and bone marrow-derived products, have emerged as potential alternatives to promote tissue healing and long-term symptom improvement.

This randomized controlled trial investigates and compares two minimally invasive orthobiologic interventions:

Bone Marrow Aspirate (BMA) - obtained from the posterior iliac crest under local anesthesia and injected into the most symptomatic region of the plantar fascia under ultrasound guidance.

Platelet-Rich Fibrin (PRF) - prepared from autologous venous blood by centrifugation without anticoagulants, forming a fibrin matrix injected into the plantar fascia under ultrasound guidance.

All procedures are performed under sterile conditions and tibial nerve regional anesthesia.

Pain and safety will be monitored using the Visual Analog Scale (VAS) and by recording adverse events at the following time points: baseline (0), 30 minutes, 1, 6, 12, and 24 months after the procedure.

Functional outcomes will be collected with Modified AOFAS Score at baseline, 1, 6, 12, and 24 months. Ultrasonography will measure plantar fascia thickness immediately before the intervention and at 12 months.

This research contributes to the growing evidence supporting orthobiologic therapies as viable, minimally invasive options for chronic plantar fasciitis management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years.
* Clinical diagnosis of chronic plantar fasciitis for more than 6 months, confirmed by ultrasonography (increased plantar fascia thickness and hypoechogenicity).
* Persistent heel pain refractory to conventional conservative treatment (stretching, orthotics, physical therapy, or corticosteroid injections).
* Visual Analog Scale (VAS) pain score ≥ 4 at baseline.
* Ability and willingness to comply with study procedures and follow-up assessments.
* Signed informed consent.

Exclusion Criteria:

* Previous foot or ankle surgery on the affected limb.
* Acute trauma, infection, or ulceration in the region of the plantar fascia.
* Systemic inflammatory diseases (e.g., rheumatoid arthritis, lupus, psoriatic arthritis).
* Metabolic or endocrine disorders interfering with healing (e.g., diabetes mellitus with poor glycemic control, thyroid disorders).
* Current use of systemic corticosteroids, immunosuppressants, or anticoagulants.
* Active neoplasia or hematologic disorders.
* Pregnancy or breastfeeding.
* Peripheral vascular disease or neuropathy affecting the lower limbs.
* Contraindications to local anesthesia or venipuncture.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity (VAS) and occurrence of adverse events | baseline (0), 30 minutes, 1, 6, 12, and 24 months
  Pain intensity measured by Visual Analog Scale (VAS) and documentation of any adverse events, assessed at each time point by a blinded evaluator.

SECONDARY OUTCOMES:
Change in Modified AOFAS Score | baseline, 1, 6, 12, 24 months
  Improvement in the American Orthopaedic Foot and Ankle Society (AOFAS) score compared to baseline, reflecting pain and function.
Change in Plantar Fascia Thickness by Ultrasound | Pre-procedure (baseline) and 12 months
  Variation in plantar fascia thickness (in millimeters) evaluated by ultrasound before the procedure and at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Fonseca, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo - Hospital São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the findings of this study will be made available upon reasonable request after publication of the main results. Data will be shared with qualified researchers for academic purposes only, upon approval by the principal investigator and the ethics committee.
Time Frame: The IPD will be available beginning 6 months after publication and for up to 3 years thereafter.
Access Criteria: Researchers must provide a methodologically sound proposal and obtain approval from the study's principal investigator (Lucas Fonseca, MD). Data access will be granted through a secure data transfer agreement.